CLINICAL TRIAL: NCT00286455
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of SYR110322 (SYR-322) Compared With Placebo in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of Alogliptin in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-PLC-010; 2005-004670-24 (EudraCT Number); U1111-1113-8462 (Registry Identifier: WHO)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alogliptin — Alogliptin 12.5 mg, tablets, orally, once daily for up to 26 weeks.
  Other Names: SYR110322; SYR-322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin — Alogliptin 25 mg, tablets, orally, once daily for up to 26 weeks.
  Other Names: SYR110322; SYR-322
  Arms: Alogliptin 25 mg QD
Drug: Placebo — Alogliptin placebo-matching tablets, orally, once daily for up to 26 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alogliptin, once daily (QD), in adults with type 2 diabetes.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% are type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

The aim of the current study is to evaluate the efficacy of alogliptin in subjects with type 2 diabetes mellitus who are inadequately controlled and who have failed treatment with diet and exercise. Individuals who participate in this study will be required to commit to a screening visit and up to 14 additional visits at the study center. Study participation is anticipated to be about 34 weeks (or 8.5 months).

ELIGIBILITY:
Inclusion Criteria

* Type 2 diabetes mellitus, experiencing inadequate glycemic control, and are receiving no current antidiabetic therapy. Subjects will qualify if both of the following conditions apply:

  * Subject has failed treatment with diet and exercise for at least one month prior to Screening
  * Subject has received less than 7 days of any antidiabetic therapy within the 3 months prior to Screening Diagnosis of type 2 diabetes must be based on current American Diabetes Association criteria.
* Body mass index greater than or equal to 23 kg/m2 and less than or equal to 45 kg/m2
* Fasting C-peptide concentration greater than or equal to 0.8 ng per mL (greater than or equal to 0.26 nmol per L). (If this screening criterion is not met, the subject still qualifies if C-peptide greater than or equal to1.5 ng per mL (greater than or equal to 0.50 nmol per L) after a challenge test.
* Glycosylated hemoglobin concentration between 7.0% and 10.0%, inclusive
* If regular use of other, non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
* Systolic blood pressure less than or equal to 180 mm Hg and diastolic pressure less than or equal to 110 mm Hg
* Hemoglobin greater than or equal to 12 g per dL (greater than or equal to 120 gm per L) for males and greater than or equal to 10 g per dL (greater than or equal to 100 gm per L) for females
* Alanine aminotransferase less than or equal to 3 times the upper limit of normal
* Serum creatinine less than or equal to 2.0 mg per dL (less than or equal to 17 micromol per L)
* Thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the subject is clinically euthyroid
* Neither pregnant (confirmed by laboratory testing in females of childbearing potential) nor lactating.
* Female subjects of childbearing potential must be practicing adequate contraception. Adequate contraception must be practiced for the duration of participation in the study.
* Able and willing to monitor their own blood glucose concentrations with a home glucose monitor.
* No major illness or debility that in the investigator's opinion prohibits the subject from completing the study.
* Able and willing to provide written informed consent.

Exclusion Criteria

* Urine albumin to creatinine ratio of greater than1000 μg per mg (greater than 113 mg per mol) at Screening. If elevated, the subject may be rescreened within 1 week.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening. (A history of treated cervical intraepithelial neoplasia 1 or cervical intraepithelial neoplasia 2 is allowed).
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* History of treated diabetic gastric paresis.
* New York Heart Association Class III or IV heart failure regardless of therapy. Currently treated subjects who are stable at Class I or II are candidates for the study.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that will affect the subject's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* History of alcohol or substance abuse within the 2 years prior to Screening.
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening.
* Prior treatment in an investigational study of alogliptin.
* Excluded Medications

  * Treatment with antidiabetic agents (other than study drug following enrollment in the study) is not allowed within the 3 months prior to Screening and through the completion of the end-of-treatment/early termination procedures. (Exception: if a subject has received other antidiabetic therapy for less than 7 days within the 3 months prior to Screening.)
  * Treatment with weight-loss drugs, any investigational antidiabetics, or oral or systemically injected glucocorticoids is not allowed from 3 months prior to randomization through the completion of the end-of-treatment/early termination procedures. Inhaled corticosteroids are allowed.
  * Subjects are not to take any medications, including over-the-counter products, without first consulting with the Study Doctor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (67):
- United States (50):
  - Birmingham, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Anaheim, California
  - Artesia, California
  - Fresno, California
  - Lafayette, California
  - Northridge, California
  - Orange, California
  - San Diego, California
  - Walnut Creek, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Cocoa Beach, Florida
  - Kissimmee, Florida
  - Longwood, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Saint Cloud, Florida
  - Honolulu, Hawaii
  - Idaho Falls, Idaho
  - Avon, Indiana
  - Elkhart, Indiana
  - Evansville, Indiana
  - Baltimore, Maryland
  - Sudbury, Massachusetts
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Burlington, North Carolina
  - Morehead City, North Carolina
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Lansdale, Pennsylvania
  - West Grove, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Cookeville, Tennessee
  - Milan, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Texarkana, Texas
  - Burlington, Vermont
- Multiple Cities, Argentina
- Multiple Cities, Australia
- Multiple Cities, Brazil
- Multiple Cities, Chile
- Multiple Cities, Czechia
- Multiple Cities, Dominican Republic
- Multiple Cities, Germany
- Multiple Cities, Guatemala
- Multiple Cities, Hungary
- Multiple Cities, India
- Multiple Cities, Mexico
- Multiple Cities, Netherlands
- Multiple Cities, New Zealand
- Multiple Cities, Peru
- Multiple Cities, Poland
- Multiple Cities, South Africa
- Multiple Cities, United Kingdom

REFERENCES:
- [Result] DeFronzo RA, Fleck PR, Wilson CA, Mekki Q; Alogliptin Study 010 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor alogliptin in patients with type 2 diabetes and inadequate glycemic control: a randomized, double-blind, placebo-controlled study. Diabetes Care. 2008 Dec;31(12):2315-7. doi: 10.2337/dc08-1035. Epub 2008 Sep 22. PMID 18809631
- [Result] Pratley RE, McCall T, Fleck PR, Wilson CA, Mekki Q. Alogliptin use in elderly people: a pooled analysis from phase 2 and 3 studies. J Am Geriatr Soc. 2009 Nov;57(11):2011-9. doi: 10.1111/j.1532-5415.2009.02484.x. Epub 2009 Sep 30. PMID 19793357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 117 investigative sites in 16 countries from 24 February 2006 to 05 July 2007.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus were enrolled in one of 3, once-daily (QD) treatment groups.
Groups:
- Placebo QD: Alogliptin placebo-matching tablets, orally, once daily for up to 26 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily for up to 26 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily for up to 26 weeks.
Period: Overall Study
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Started | 65 | 133 | 131
Completed | 40 | 105 | 107
Not Completed | 25 | 28 | 24
Not completed — Hyperglycemia rescue | 19 | 13 | 10
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 3 | 3
Not completed — Physician Decision | 3 | 0 | 2
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Participant Non-compliance | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Total
Number analyzed (Participants) | 65 | 133 | 131 | 329
Age, Customized [Number; unit: participants]
  <65 years | 53 | 110 | 111 | 274
  Between 65 and 74 years | 8 | 18 | 16 | 42
  ≥75 years | 4 | 5 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 68 | 54 | 154
  Male | 33 | 65 | 77 | 175

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 26 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at the week 26 visit. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 131 | 128
percentage of Glycosylated Hemoglobin | -0.02 (0.094) | -0.56 (0.065) | -0.59 (0.066)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Null Hypothesis: No difference between treatment and placebo arms in change from baseline in glycosylated hemoglobin. Sample size calculated based on normally distributed means. For comparison of either dose vs. placebo (2-sample t-test), study sample size >=325 subjects had 95% power to detect a treatment difference as small as 0.5% in the supportive per protocol analysis set assuming SD=0.8%, 2-sided >0.05 significance level and >=80% of subjects meeting per protocol criteria; Test type: Superiority or Other; p < 0.001, ANCOVA — A step-down strategy was used for the primary analysis. First, the 25mg dose was compared to placebo at the 2-sided 0.05 significance level. The 12.5 mg dose was compared to placebo only if the comparison of the 25mg dose to placebo was significant; Treatment and geographic region as class variables; diabetes duration and baseline value for the endpoint (HbA1c) as covariates; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.76 to -0.31] — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.80 to -0.35] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF). Smaller "n" at earlier timepoints due to unavailable prior values to carry forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 123 | 120
percentage of Glycosylated Hemoglobin | -0.11 (0.052) | -0.37 (0.035) | -0.45 (0.036)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; Treatment and geographic region as class variables; diabetes duration and baseline value for the endpoint parameter as covariates; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.39 to -0.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.46 to -0.21] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 131 | 128
percentage of Glycosylated Hemoglobin | -0.13 (0.072) | -0.53 (0.049) | -0.64 (0.050)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.57 to -0.23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.68 to -0.33] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 131 | 128
percentage of Glycosylated Hemoglobin | -0.13 (0.080) | -0.57 (0.055) | -0.66 (0.056)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-0.63 to -0.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.73 to -0.35] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 131 | 128
percentage of Glycosylated Hemoglobin | -0.12 (0.085) | -0.59 (0.058) | -0.65 (0.059)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.68 to -0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.74 to -0.33] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 131 | 128
percentage of Glycosylated Hemoglobin | -0.12 (0.090) | -0.58 (0.062) | -0.61 (0.062)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.67 to -0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.70 to -0.27] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 1).
Description: The change between the value of fasting plasma glucose collected at final visit or week 1 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 1.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 60 | 120 | 121
mg/dL | 4.6 (3.45) | -8.6 (2.41) | -14.0 (2.41)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -13.2, 95% CI 2-sided [-21.5 to -5.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -18.7, 95% CI 2-sided [-27.0 to -10.4] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 62 | 129 | 126
mg/dL | 3.8 (3.47) | -14.6 (2.38) | -17.6 (2.42)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -18.4, 95% CI 2-sided [-26.7 to -10.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -21.4, 95% CI 2-sided [-29.7 to -13.0] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 131 | 129
mg/dL | 2.8 (3.63) | -15.6 (2.51) | -21.6 (2.54)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -18.4, 95% CI 2-sided [-27.1 to -9.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -24.4, 95% CI 2-sided [-33.2 to -15.7] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 131 | 129
mg/dL | 2.5 (4.20) | -14.3 (2.91) | -19.8 (2.94)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -16.7, 95% CI 2-sided [-26.8 to -6.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -22.3, 95% CI 2-sided [-32.4 to -12.2] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 132 | 129
mg/dL | 1.2 (4.29) | -15.3 (2.97) | -20.0 (3.01)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -16.5, 95% CI 2-sided [-26.8 to -6.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -21.2, 95% CI 2-sided [-31.6 to -10.8] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 132 | 129
mg/dL | 5.2 (4.64) | -14.6 (3.21) | -18.2 (3.25)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -19.8, 95% CI 2-sided [-30.9 to -8.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -23.4, 95% CI 2-sided [-34.6 to -12.2] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 132 | 129
mg/dL | 7.0 (4.73) | -12.3 (3.27) | -17.3 (3.31)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -19.3, 95% CI 2-sided [-30.6 to -8.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -24.3, 95% CI 2-sided [-35.7 to -12.9] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 26).
Description: The change between the value of fasting plasma glucose collected at week 26 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 132 | 131
mg/dL | 11.3 (5.24) | -10.3 (3.62) | -16.4 (3.67)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -21.6, 95% CI 2-sided [-34.1 to -9.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -27.8, 95% CI 2-sided [-40.4 to -15.1] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With Marked Hyperglycemia (Fasting Plasma Glucose ≥ 200 mg Per dL).
Description: The number of participants with a fasting plasma glucose value greater than or equal to 200 mg per dL at any measurement time point during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set)and had at least 1 post-baseline FPG measurement.
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 130
participants | 30 | 44 | 33
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.165, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 0.569, 95% CI 2-sided [0.257 to 1.262] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.008, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 0.320, 95% CI 2-sided [0.138 to 0.739] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

16. Secondary Outcome: Number of Participants Requiring Rescue.
Description: The number of participants requiring rescue for failing to achieve pre-specified glycemic targets during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 19 | 13 | 10
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 0.194, 95% CI 2-sided [0.073 to 0.516] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 0.145, 95% CI 2-sided [0.052 to 0.405] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

17. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 4).
Description: The change between the value of fasting proinsulin collected at week 4 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 57 | 118 | 117
pmol/L | 2.9 (3.24) | -4.7 (2.22) | -10.4 (2.24)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.056, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-15.3 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -13.3, 95% CI 2-sided [-21.1 to -5.5] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 8).
Description: The change between the value of fasting proinsulin collected at week 8 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 128 | 124
pmol/L | -3.9 (3.60) | -3.1 (2.46) | -1.4 (2.51)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.850, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-7.8 to 9.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.571, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-6.2 to 11.2] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 12).
Description: The change between the value of fasting proinsulin collected at week 12 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 129 | 124
pmol/L | -2.8 (3.10) | -3.2 (2.11) | -8.5 (2.16)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.917, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-7.8 to 7.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.133, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-13.2 to 1.7] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 16).
Description: The change between the value of fasting proinsulin collected at week 16 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 129 | 124
pmol/L | -0.6 (3.42) | -4.5 (2.33) | -6.6 (2.38)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.348, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-12.1 to 4.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.152, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-14.3 to 2.2] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 20).
Description: The change between the value of fasting proinsulin collected at week 20 and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 129 | 124
pmol/L | -0.8 (2.75) | -6.0 (1.87) | -6.3 (1.91)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.120, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-11.7 to 1.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.104, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-12.1 to 1.1] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in Fasting Proinsulin (Week 26).
Description: The change between the value of fasting proinsulin collected at week 26 or final visit and fasting proinsulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 129 | 124
pmol/L | -2.1 (2.87) | -6.1 (1.96) | -7.4 (2.00)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.247, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-10.9 to 2.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.129, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-12.3 to 1.6] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Change From Baseline in Insulin (Week 4).
Description: The change between the value of insulin collected at week 4 and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 55 | 118 | 117
ϻIU/mL | 0.87 (1.430) | 0.14 (0.965) | -1.27 (0.973)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.671, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-4.14 to 2.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.218, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-5.57 to 1.27] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Change From Baseline in Insulin (Week 8).
Description: The change between the value of insulin collected at week 8 and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 128 | 124
ϻIU/mL | -0.35 (1.520) | 1.18 (1.023) | 0.94 (1.042)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.403, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.54, 95% CI 2-sided [-2.07 to 5.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.487, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-2.35 to 4.93] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Change From Baseline in Insulin (Week 12).
Description: The change between the value of insulin collected at week 12 and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ϻIU/mL | -1.66 (1.467) | 0.94 (0.984) | -1.60 (1.006)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.143, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.60, 95% CI 2-sided [-0.88 to 6.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.974, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-3.46 to 3.57] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Change From Baseline in Insulin (Week 16).
Description: The change between the value of insulin collected at week 16 and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ϻIU/mL | -0.41 (1.577) | 0.55 (1.058) | -1.46 (1.082)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.612, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.97, 95% CI 2-sided [-2.78 to 4.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.587, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.04, 95% CI 2-sided [-4.82 to 2.74] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Change From Baseline in Insulin (Week 20).
Description: The change between the value of insulin collected at week 20 and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ϻIU/mL | -1.32 (1.264) | -0.32 (0.847) | -1.12 (0.867)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.514, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-2.00 to 3.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.899, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-2.83 to 3.22] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Change From Baseline in Insulin (Week 26).
Description: The change between the value of insulin collected at week 26 and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ϻIU/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ϻIU/mL | -1.17 (1.404) | -0.92 (0.942) | -1.08 (0.963)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.885, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-3.09 to 3.58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.958, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-3.28 to 3.46] — [estimate comment as in outcome 1, analysis 1]

29. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 4).
Description: The change between the ratio value of proinsulin and insulin collected at week 4 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 55 | 118 | 117
ratio | 0.008 (0.0140) | -0.043 (0.0094) | -0.063 (0.0095)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.084 to -0.018] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.072, 95% CI 2-sided [-0.105 to -0.038] — [estimate comment as in outcome 1, analysis 1]

30. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 8).
Description: The change between the ratio value of proinsulin and insulin collected at week 8 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 128 | 124
ratio | 0.014 (0.0130) | -0.054 (0.0087) | -0.038 (0.0089)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.069, 95% CI 2-sided [-0.099 to -0.038] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.052, 95% CI 2-sided [-0.083 to -0.021] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 12).
Description: The change between the ratio value of proinsulin and insulin collected at week 12 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ratio | 0.025 (0.0150) | -0.043 (0.0100) | -0.047 (0.0103)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.068, 95% CI 2-sided [-0.103 to -0.032] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.073, 95% CI 2-sided [-0.109 to -0.037] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 16).
Description: The change between the ratio value of proinsulin and insulin collected at week 16 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ratio | 0.001 (0.0162) | -0.044 (0.0109) | -0.039 (0.0111)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.021, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.084 to -0.007] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.043, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.040, 95% CI 2-sided [-0.079 to -0.001] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 20).
Description: The change between the ratio value of proinsulin and insulin collected at week 20 and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ratio | 0.119 (0.0393) | -0.043 (0.0263) | -0.040 (0.0270)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.162, 95% CI 2-sided [-0.255 to -0.069] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.159, 95% CI 2-sided [-0.254 to -0.065] — [estimate comment as in outcome 1, analysis 1]

34. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio (Week 26).
Description: The change between the ratio value of proinsulin and insulin collected at week 26 or final visit and the ratio value of proinsulin and insulin collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 129 | 124
ratio | 0.046 (0.0219) | -0.040 (0.0147) | -0.038 (0.0150)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.086, 95% CI 2-sided [-0.138 to -0.034] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-0.137 to -0.032] — [estimate comment as in outcome 1, analysis 1]

35. Secondary Outcome: Change From Baseline in C-peptide (Week 4).
Description: The change between the value of C-peptide collected at week 4 and C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 59 | 119 | 120
ng/mL | 0.242 (0.1467) | 0.026 (0.1024) | 0.088 (0.1023)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.230, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.216, 95% CI 2-sided [-0.568 to 0.137] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.393, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.154, 95% CI 2-sided [-0.508 to 0.200] — [estimate comment as in outcome 1, analysis 1]

36. Secondary Outcome: Change From Baseline in C-peptide (Week 8).
Description: The change between the value of C-peptide collected at week 8 and C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 129 | 127
ng/mL | -0.014 (0.1801) | 0.070 (0.1249) | 0.269 (0.1263)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.703, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.084, 95% CI 2-sided [-0.348 to 0.515] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.203, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.282, 95% CI 2-sided [-0.153 to 0.717] — [estimate comment as in outcome 1, analysis 1]

37. Secondary Outcome: Change From Baseline in C-peptide (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 130 | 127
ng/mL | -0.104 (0.1673) | 0.064 (0.1156) | -0.091 (0.1173)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.408, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.169, 95% CI 2-sided [-0.232 to 0.569] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.949, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.391 to 0.417] — [estimate comment as in outcome 1, analysis 1]

38. Secondary Outcome: Change From Baseline in C-peptide (Week 16).
Description: The change between the value of C-peptide collected at week 16 and C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 130 | 127
ng/mL | -0.030 (0.1712) | -0.060 (0.1183) | -0.127 (0.1200)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.886, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.440 to 0.380] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.645, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.097, 95% CI 2-sided [-0.510 to 0.317] — [estimate comment as in outcome 1, analysis 1]

39. Secondary Outcome: Change From Baseline in C-peptide (Week 20).
Description: The change between the value of C-peptide collected at week 20 and C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 130 | 127
ng/mL | -0.194 (0.1288) | -0.264 (0.0890) | -0.231 (0.0903)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.656, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.070, 95% CI 2-sided [-0.378 to 0.239] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.819, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.036, 95% CI 2-sided [-0.347 to 0.275] — [estimate comment as in outcome 1, analysis 1]

40. Secondary Outcome: Change From Baseline in C-peptide (Week 26).
Description: The change between the value of C-peptide collected at week 26 or final visit and C-peptide collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 130 | 127
ng/mL | -0.282 (0.1387) | -0.360 (0.0958) | -0.279 (0.0973)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.642, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.079, 95% CI 2-sided [-0.411 to 0.253] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.986, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.332 to 0.338] — [estimate comment as in outcome 1, analysis 1]

41. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 6.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 6.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 7 | 23 | 27
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.305, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 1.686, 95% CI 2-sided [0.622 to 4.571] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.091, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 2.349, 95% CI 2-sided [0.873 to 6.321] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

42. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.0%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 15 | 63 | 58
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 3.704, 95% CI 2-sided [1.694 to 8.100] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.003, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 3.305, 95% CI 2-sided [1.505 to 7.255] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

43. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 25 | 81 | 88
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.006, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 2.905, 95% CI 2-sided [1.359 to 6.210] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 4.552, 95% CI 2-sided [2.068 to 10.017] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

44. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 0.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 0.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 19 | 67 | 72
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.004, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 2.663, 95% CI 2-sided [1.367 to 5.188] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 3.277, 95% CI 2-sided [1.671 to 6.429] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

45. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 7 | 38 | 39
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.002, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 4.331, 95% CI 2-sided [1.714 to 10.947] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.001, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 4.732, 95% CI 2-sided [1.862 to 12.025] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

46. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 3 | 11 | 16
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.153, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 2.766, 95% CI 2-sided [0.685 to 11.160] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.029, Regression, Logistic; Logistic regression model includes effects for treatment, geographic region, diabetes duration and baseline HbA1c; Odds Ratio (OR) = 4.632, 95% CI 2-sided [1.169 to 18.354] — Odd's Ratio (OR) compares alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

47. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 2.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 2.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set).
Measure: Number; unit: participants
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 64 | 133 | 131
participants | 1 | 3 | 6
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.102, Mantel Haenszel — No multiplicity adjustments; Odd's Ratio and 95% CI not estimable using logistic regression model. Tested using extended Mantel-Haenszel test
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.063, Mantel Haenszel — No multiplicity adjustments; Odd's Ratio and 95% CI not estimable using logistic regression model. Tested using extended Mantel-Haenszel test

48. Secondary Outcome: Change From Baseline in Body Weight (Week 8).
Description: The change between Body Weight measured at week 8 and Body Weight measured at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF). Smaller "n" at earlier timepoint due to unavailable prior values to carry forward
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 61 | 126 | 123
kg | -0.36 (0.232) | 0.01 (0.160) | -0.03 (0.162)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.186, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-0.18 to 0.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.237, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.22 to 0.89] — [estimate comment as in outcome 1, analysis 1]

49. Secondary Outcome: Change From Baseline in Body Weight (Week 12).
Description: The change between Body Weight measured at week 12 and Body Weight measured at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 126 | 125
kg | -0.25 (0.257) | -0.37 (0.180) | 0.05 (0.181)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.702, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.74 to 0.50] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.338, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.32 to 0.93] — [estimate comment as in outcome 1, analysis 1]

50. Secondary Outcome: Change From Baseline in Body Weight (Week 20).
Description: The change between Body Weight measured at week 20 and Body Weight measured at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 126 | 125
kg | -0.17 (0.305) | -0.18 (0.213) | -0.17 (0.215)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.978, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.74 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.991, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.73 to 0.74] — [estimate comment as in outcome 1, analysis 1]

51. Secondary Outcome: Change From Baseline in Body Weight (Week 26).
Description: The change between Body Weight measured at week 26 or final visit and Body Weight measured at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 63 | 126 | 125
kg | 0.18 (0.368) | -0.09 (0.258) | -0.22 (0.259)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.539, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.16 to 0.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.379, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.29 to 0.49] — [estimate comment as in outcome 1, analysis 1]

52. Secondary Outcome: Change From Baseline in Glucagon (Week 4).
Description: The change between the value of glucagon collected at week 4 and glucagon collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 45 | 101 | 91
pg/mL | 2.1 (2.51) | 3.6 (1.65) | 1.8 (1.75)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.616, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [-4.4 to 7.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.930, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-6.4 to 5.8] — [estimate comment as in outcome 1, analysis 1]

53. Secondary Outcome: Change From Baseline in Glucagon (Week 8).
Description: The change between the value of glucagon collected at week 8 and glucagon collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized participants who received at least one dose of study drug (Full Analysis Set), and who had measurements at baseline and at the visit. Missing data are imputed using last observation carried forward (LOCF).) Smaller "n" at earlier timepoints due to unavailable prior values to carry forward.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 50 | 109 | 100
pg/mL | -1.2 (2.38) | -0.9 (1.59) | -0.2 (1.66)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.915, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-5.3 to 6.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.745, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-4.8 to 6.7] — [estimate comment as in outcome 1, analysis 1]

54. Secondary Outcome: Change From Baseline in Glucagon (Week 12).
Description: The change between the value of glucagon collected at week 12 and glucagon collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 50 | 111 | 101
pg/mL | -1.2 (2.30) | 0.8 (1.52) | 2.8 (1.60)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.466, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-3.4 to 7.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.154, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-1.5 to 9.6] — [estimate comment as in outcome 1, analysis 1]

55. Secondary Outcome: Change From Baseline in Glucagon (Week 16).
Description: The change between the value of glucagon collected at week 16 and glucagon collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 50 | 111 | 101
pg/mL | 2.4 (2.53) | 3.3 (1.67) | 3.4 (1.76)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.774, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-5.1 to 6.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.761, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-5.2 to 7.1] — [estimate comment as in outcome 1, analysis 1]

56. Secondary Outcome: Change From Baseline in Glucagon (Week 20).
Description: The change between the value of glucagon collected at week 20 and glucagon collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 50 | 111 | 101
pg/mL | 1.6 (2.50) | 3.3 (1.65) | 3.5 (1.74)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.559, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-4.2 to 7.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.523, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-4.1 to 8.0] — [estimate comment as in outcome 1, analysis 1]

57. Secondary Outcome: Change From Baseline in Glucagon (Week 26).
Description: The change between the value of glucagon collected at week 26 or final visit and glucagon collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 50 | 111 | 101
pg/mL | 5.2 (2.66) | 4.2 (1.76) | 2.4 (1.85)
Statistical Analysis 1: Comparison: Placebo QD vs Alogliptin 12.5 mg QD; Test type: Superiority or Other; p = 0.739, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-7.4 to 5.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo QD vs Alogliptin 25 mg QD; Test type: Superiority or Other; p = 0.388, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-9.3 to 3.6] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious event) after the last dose of double-blind drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo QD | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Serious Adverse Events (participants affected / at risk) | 2/64 | 5/133 | 1/132
Other Adverse Events (participants affected / at risk) | 32/64 | 48/133 | 39/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=64) | Alogliptin 12.5 mg QD (N=133) | Alogliptin 25 mg QD (N=132)
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Noncardiac chest pain (General disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=64) | Alogliptin 12.5 mg QD (N=133) | Alogliptin 25 mg QD (N=132)
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 6
Nasopharyngitis (Infections and infestations) | 5 | 12 | 10
Headache (Nervous system disorders) | 3 | 10 | 9
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 2
Urinary tract infection (Infections and infestations) | 3 | 7 | 5
Dizziness (Nervous system disorders) | 3 | 4 | 2
Hypertension (Vascular disorders) | 1 | 4 | 5
Pharyngitis (Infections and infestations) | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Blister (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2
Sinusitis (Infections and infestations) | 2 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.